CLINICAL TRIAL: NCT01221194
Title: Therapeutic Stockings to Prevent Foot Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Larry Lavery, Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STU 082010-090
Record Dates: First submitted 2010-10-13; First posted 2010-10-14 (Estimated); Results first posted 2020-08-26 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Diabetes
Keywords: diabetes; foot ulcer prevention; therapeutic stockings
MeSH Terms: conditions — Diabetes Mellitus | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Standard therapy (Active Comparator): Standard therapy consisting of education, regular foot care and protective shoes and insoles. The standard therapy group will use the stockings they normally wear.
  Interventions: Behavioral: Standard therapy
- PFC Stockings (Active Comparator): The stocking therapy group will be given PFC shear reducing stockings to wear.
  Interventions: Device: PFC Stockings

INTERVENTIONS:
Behavioral: Standard therapy — Standard therapy consisting of education, regular foot care and protective shoes and insoles. The standard therapy group will use the stockings they normally wear.
  Arms: Standard therapy
Device: PFC Stockings — A pressure and friction reducing stocking. The novelty of the PFC Sock stems from its innovative double layer structure and technological fibre composition. These simultaneously and significantly reduce both pressure and friction in a format that is practical for everyday wear with therapeutic shoes in high-risk cases.
  Arms: PFC Stockings

SUMMARY:
1. To evaluate the efficacy of a therapeutic stockings (Protective Foot Care stockings, PFC) in reducing the incidence of diabetic foot pathology among high-risk patients.
2. To evaluate perceived health-related quality of life as compared to guideline directed usual care in patients who use the PFC stockings.

DETAILED DESCRIPTION:
We will identify a cohort of high-risk diabetic patients and assign them to two treatment groups. We plan to enroll patients from three sites: Scott and White Hospital in Temple Texas, Manchester Royal Infirmary, UK , and Trinity College Dublin at St James Hospital.. The two treatment arms will involve a Standard Therapy Group, and a Stocking Therapy Group. The Stocking Therapy group will use the special padded and friction reducing stockings in their standard shoes during the course of the study. Patient enrollment will occur over a one-year period. All patients will be followed for 30 months. The Standard Therapy Group will receive therapeutic shoes, standard insoles, patient education and regular foot evaluations by a physician every 10-12 weeks. The Stocking Therapy Group will receive standard therapy as described above but use the special stockings instead of their usual hose. The investigator at each site will be blinded regarding the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Men or women 18 years old or older
* Diagnosis of Diabetes Mellitus*
* History of diabetes related foot ulceration

Spanish-speaking subjects will be eligible to participate.

Exclusion Criteria:

* Active Charcot Arthropathy
* Gangrene, active infection
* Midfoot or higher level amputation
* Alcohol or substance abuse within 6 months
* Unreliable, unwilling or unable to comprehend informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 381 (Actual)
Dates: Start 2010-10; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Lavery, DPM, Principal Investigator — UT Southwestern Medical Center at Dallas
Locations (4):
- United States (3):
  - Parkland Health & Hospital Systems, Dallas, Texas
  - UT Southwestern Medical Center at Dallas, Dallas, Texas
  - Scott & White, Temple, Texas
- University of Manchester, Manchester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PFC Stockings | Standard Therapy
Started | 195 | 186
Completed | 195 | 186
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PFC Stockings | Standard Therapy | Total
Number analyzed (Participants) | 195 | 186 | 381
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.06 (11.14) | 56.08 (6.76) | 53.72 (9.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 43 | 94
  Male | 144 | 143 | 287
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 56 | 42 | 98
  Not Hispanic or Latino | 133 | 136 | 269
  Unknown or Not Reported | 6 | 8 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 13 | 19
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 23 | 40
  White | 166 | 144 | 310
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 125 | 109 | 234
  United Kingdom | 70 | 77 | 147

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Developed Foot Ulcer During Study Time Frame
Description: An ulceration will be defined as full thickness loss of epidermis and dermis or involvement of deeper structures.
Time Frame: 30 months
Measure: Count of Participants; unit: Participants
Arm/Group | PFC Stockings | Standard Therapy
Number analyzed (Participants) | 195 | 186
Participants | 76 | 82

ADVERSE EVENTS:
Arm/Group | PFC Stockings | Standard Therapy
All-Cause Mortality (participants affected / at risk) | 7/195 | 7/186
Serious Adverse Events (participants affected / at risk) | 30/195 | 16/186
Other Adverse Events (participants affected / at risk) | 99/195 | 99/186
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PFC Stockings (N=195) | Standard Therapy (N=186)
Foot related readmission (Infections and infestations) | 13 (16) | 6 (7)
Non-foot related hospitalization (Musculoskeletal and connective tissue disorders) | 17 (22) | 10 (12)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PFC Stockings (N=195) | Standard Therapy (N=186)
Osteomyelitis (Infections and infestations) | 1 | 4
Amputation (Surgical and medical procedures) | 18 | 9
New foot ulcer (Skin and subcutaneous tissue disorders) | 76 | 82
Mechanical fall (Nervous system disorders) | 2 (2) | 2 (2)
Foot fracture (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No